CLINICAL TRIAL: NCT05242523
Title: Automated Stress Detection and Restoration in Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Southern California NIOSH Education and Research Center (Unknown)
Responsible Party: Principal Investigator, Burcin Becerik-Gerber, Professor, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: UP-21-00484
Record Dates: First submitted 2022-01-20; First posted 2022-02-16 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No exposure to smells.
- Olfactory Condition - 1 (Experimental): Participants in this condition will be exposed to the smell of natural wood scent continuously. A diffuser with essential oils will be turned on during that time to deliver the smell.
  Interventions: Other: Natural wood scent
- Olfactory Condition - 2 (Experimental): Participants in this condition will be exposed to the smell of Bergamot scent continuously. A diffuser with essential oils will be turned on during that time to deliver the smell.
  Interventions: Other: Bergamot scent

INTERVENTIONS:
Other: Bergamot scent — The scent of bergamot is fruity and citrusy, with floral hints and spice notes.
  Arms: Olfactory Condition - 2
Other: Natural wood scent — Wood notes tend to be rich and warm, often forming the base of a scent due to their aromatic weight.
  Arms: Olfactory Condition - 1

SUMMARY:
This study aims at establishing a laboratory experiment that mimics office work stressors, examining the feasibility of automated stress detection, and identifying the most significant physiological and/or behavioral features that can be used to differentiate between positive stress (eustress) and negative stress (distress). Additionally, we will investigate if triggering the olfactory (exposing participants to pleasant smells) senses would help reduce stress.

DETAILED DESCRIPTION:
The experiment is divided into 2 main phases:

The first phase is the eustress-distress data collection: In this phase, participants will complete three conditions:

1. "No-stress": Participants will sit idle on their desks without performing any task. This is important to record a baseline of physiological signals that will allow us to compare the physiological responses in later stages.
2. "Low-stress work": Participants will be asked to prepare a brief presentation about a familiar topic (e.g., favorite types of food, TV shows, academic work). A strict time limit will not be provided; instead, participants will be told that they have at least 30 minutes and up to 40 minutes if they need that amount of time to complete the presentation.
3. "High-stress work": Participants will be required to prepare a presentation about an unfamiliar topic with a time limit of 30 minutes. The topic and the requirements will be carefully established to make the completion of the presentation achievable but at the same time to create a sense of time pressure, heavy workload, and unfamiliarity with the task. We will employ a concept similar to the Trier Social Stress Test, in which participants are required to develop and deliver a speech to a panel. This test has been employed in several studies as a means of inducing high-stress reactions. In our study, participants will be informed that a two-person judging committee will be scoring their work performance by watching through a Zoom shared screen. Participants will be told that their final score will be compared to all other study participants such that the highest scoring individuals will receive an award. The committee's "score" will be presented on the screen beginning at 100 and will be decreased and increased in a standardized manner across all participants. Changes in the score will appear at uneven intervals such that the participants do not recognize a pattern but associate the scoring with the judging committee noticing some sort of work flaw or issue. A countdown clock with time remaining will be presented on the screen, recorded office noise (e.g., printers, distant chatting, computers) will be played in the background, and temperature will be increased outside the comfort range. In addition, participants will be subject to interruptions including pop-up messages, calls or emails every 5 minutes to ask about progress.

During the three conditions (idle, low stress, high stress) participants will be asked 5 questions every 5 minutes:

1. In the last five minutes, to what extent did you consider the work you are performing as an opportunity or challenge?
2. In the last five minutes, to what extent did you consider the work you are performing as a source of pressure?
3. Over the last five minutes, how would you rate your productivity?
4. Over the last five minutes, how would you rate your mood?
5. Over the last five minutes, how would you rate your stress level?

The second phase is meant to investigate if triggering the olfactory (exposing participants to pleasant smells) senses would help reduce stress.

For that, participants will be given a task that an office worker usually conducts in their everyday work (e.g., typing a paragraph in a word document, organizing a spreadsheet) for 20 minutes. During the 20 minutes, participants will get exposed to one of the following three conditions:

1. Control group - 20 participants: No exposure to smells or change in office light settings.
2. Olfactory group 1 - 20 participants: No change in office light settings, but participants in this condition will be exposed to the smell of natural wood scent continuously. A diffuser with essential oils will be turned on during that time to deliver the smell.
3. Olfactory group 2 - 20 participants: No change in office light settings, but participants in this condition will be exposed to the smell of Bergamot scent continuously. A diffuser with essential oils will be turned on during that time to deliver the smell.

Following this, participants will be asked to rate their anxiety/stress levels using the state anxiety trait survey and how they perceived the exposure to the scents.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be older than 18.
2. Participants should be proficient at speaking and writing in English.
3. Qualified participants should have a normal or corrected-to-normal vision, and a normal sense of smell.

Exclusion Criteria:

1. Participants will be screened to make sure that they don't have any physical or psychological-related problems that make them sensitive to stress-inducing tasks.
2. Participants who are taking any medication to regulate their blood pressure will not be allowed to participate in the study as these medications might affect the quality of the blood volume pulse-related data.
3. Pregnant women are not allowed to participate in this study.
4. Participants using prescription medication, diagnosed with color blindness, rhinitis, or hay fever, or have allergic reactions to essential oils ( e.g., contact dermatitis, allergic rhinitis) will not be allowed to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Heart rate | Throughout study participation, up to 120 minutes
  Heart rate will be collected through a sensor attached to the participant's chest at a collection rate of 1 heart rate reading per second. The average heart rate will be examined across study conditions.
Electrodermal activity | Throughout study participation, up to 120 minutes
  Electrodermal activity will be collected through a sensor placed on the wrist similar to a watch, with data collection at a rate of 4 readings per second. The average electrodermal activity will be examined across study conditions.
Blink rate | Throughout study participation, up to 120 minutes
  A facial detection algorithm will be used to detect the blinking rate of the participant from a camera that collects 10 frames per second. The average blink rate will be examined across study conditions.
Gaze angle | Throughout study participation, up to 120 minutes
  A facial detection algorithm will be used to detect the gaze angle direction of the participant from a camera that collects 10 frames per second. The durations of gaze angles will be examined across study conditions.

SECONDARY OUTCOMES:
Mouse clicks | Throughout study participation, up to 120 minutes
  The number of mouse clicks will be recorded using a logger software installed on the computer. The frequency of mouse clicks will be examined across study conditions.
Keyboard keystrokes | Throughout study participation, up to 120 minutes
  The number of keystrokes will be recorded using a logger software installed on the computer. The frequency of keystrokes will be examined across study conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Burcin Becerik-Gerber, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No